CLINICAL TRIAL: NCT00727402
Title: The Longitudinal Evaluation of Silicone Hydrogel (LASH) Contact Lens Study
Brief Title: Longitudinal Evaluation of Silicone Hydrogel (LASH) Study
Acronym: LASH
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Loretta Szczotka-Flynn, Professor, Case Western Reserve University
Other Study IDs: K23EY015270-01 (NIH)
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Results first posted 2011-02-10 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Corneal Infiltrates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tear samples contact lenses bacteria isolated from contact lenses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: healthy patients fit into lotrafilcon A contact lenses for continuous wear

SUMMARY:
The LASH Contact Lens Study is a prospective longitudinal study of silicone hydrogel (SH) contact lens wearers who sleep in their lenses for up to 29 consecutive nights (30 days) of continuous wear (CW), with monthly disposal. Up to 207 healthy nearsighted or farsighted patients with minimal or no astigmatism and no contraindications to CW lens use will be followed for 1 year. The primary outcome measure is the time to development of a corneal inflammatory event (CIE) as defined by slit lamp findings and patient symptoms. The main exposure of interest is corneal staining. Other key exploratory variables include bacterial contamination of study lenses and inflammatory mediators found in the tear film.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 15 years old. Children younger than this may not be mature enough for CW, and may have difficulty following the strict instructions required for CW or sitting through the exam procedures.
2. The patient must have clear central corneas and free of any anterior segment disorders.
3. The patient must have a spectacle corrected spherical refractive error between +5.50 D and -11.00 D with less than or equal to 1.00 D refractive cylinder. The parameters of the Ciba Vision Night and Day Lenses range from +6.00 to -10.00 D, and can correct the refractive range of this population. Monovision correction will be allowed only if the near eye does not exceed +6.00 D.
4. The patient must be correctable to 20/25 or better with spectacles. Amblyopia will be excluded.
5. Flat and steep corneal curvatures from SimK readings must be between 39.00 and 48.00 D. Corneal curvatures outside this range may be indicative of a disease state, and patients are not expected to comfortably wear either the 8.4 mm or 8.6 mm base curve available in Night and Day.(Dumbleton K 2002)
6. Can be successfully fit with lotrafilcon A lenses at the enrollment visit.

Exclusion Criteria:

1. The patient has worn rigid gas permeable lenses within the last 30 days or PMMA lenses within the last 3 months. These lenses can transiently alter the corneal shape and influence the fitting of soft lenses.
2. The patient must not be a current extended wear user of lotrafilcon A lenses.
3. The patient has an autoimmune disease (except for Hashimoto's Thyroiditis), immunocompromising disease, connective tissue disease, atopic dermatitis, insulin dependent diabetes, or any other systemic disease that in the investigator's opinion will affect ocular health.
4. The patient is taking chronic systemic medications such as corticosteroids, antimetabolites, or non-steroidal anti-inflammatory agents or any other medication that in the investigator's opinion will affect ocular physiology.
5. The patient has any ocular disease or condition such as aphakia, corneal dystrophies, corneal edema, external ocular infection, iritis, or had any anterior segment surgery.
6. The patient is taking any ocular medications.
7. The patient must have less than or equal to grade 2 on any of the slit lamp observations of: upper tarsal papilla, corneal staining, corneal neovascularization, conjunctival injection, and lid erythema or scales. Slit lamp findings higher than grade 2 bias the patient toward an adverse event and it may be difficult to detect true change related to CW.
8. The patient is pregnant.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: study volunteers from academic community willing to wear extended wear contact lenses
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2006-10; Primary Completion 2009-01 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loretta B Szczotka-Flynn, OD, MS, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Szczotka-Flynn L, Lass JH, Sethi A, Debanne S, Benetz BA, Albright M, Gillespie B, Kuo J, Jacobs MR, Rimm A. Risk factors for corneal infiltrative events during continuous wear of silicone hydrogel contact lenses. Invest Ophthalmol Vis Sci. 2010 Nov;51(11):5421-30. doi: 10.1167/iovs.10-5456. Epub 2010 Jun 10. PMID 20538985
- [Result] Szczotka-Flynn LB, Bajaksouzian S, Jacobs MR, Rimm A. Risk factors for contact lens bacterial contamination during continuous wear. Optom Vis Sci. 2009 Nov;86(11):1216-26. doi: 10.1097/OPX.0b013e3181bbca18. PMID 19786927
- [Result] Szczotka-Flynn L, Benetz BA, Lass J, Albright M, Gillespie B, Kuo J, Fonn D, Sethi A, Rimm A. The association between mucin balls and corneal infiltrative events during extended contact lens wear. Cornea. 2011 May;30(5):535-42. doi: 10.1097/ICO.0b013e3181fb8644. PMID 21173699
- [Derived] Tagliaferri A, Love TE, Szczotka-Flynn LB. Risk factors for contact lens-induced papillary conjunctivitis associated with silicone hydrogel contact lens wear. Eye Contact Lens. 2014 May;40(3):117-22. doi: 10.1097/ICL.0000000000000019. PMID 24681609

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observational
Started | 205
Completed | 89
Not Completed | 116
Not completed — Physician Decision | 116

BASELINE CHARACTERISTICS:
Arm/Group | Observational
Number analyzed (Participants) | 205
Age Continuous [Mean (Standard Deviation); unit: years] | 32.8 (5)
Age, Customized [Number; unit: participants]
  <=21 years | 26
  Between 21 and 50 years | 163
  >50 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157
  Male | 48
Region of Enrollment [Number; unit: participants]
  United States | 205

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Corneal Inflammatory Events
Description: Unadjusted cumulative incidence of corneal inflammatory events (CIE)using survival analysis methods. CIE are corneal infiltrates found in an otherwise clear cornea.
Time Frame: annual
Measure: Mean (95% Confidence Interval); unit: annual incidence per 100 subjects
Units Other Than Participants: eyes
Arm/Group | Observational
Number analyzed (Participants) | 205
Number analyzed (eyes) | 410
annual incidence per 100 subjects | 26.7 [20.1 to 35.0]

ADVERSE EVENTS:
Arm/Group | Observational
Serious Adverse Events (participants affected / at risk) | 0/205
Other Adverse Events (participants affected / at risk) | 58/205
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational (N=205)
corneal inflammatory event (Eye disorders) | 38 (44)
Other non-Corneal Inflammatory Event (Eye disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No